CLINICAL TRIAL: NCT04449692
Title: Low-dose Dasiglucagon for Prevention of Insulin-Induced Hypoglycemia in People With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-20013256; 2020-000551-12 (EudraCT Number); H-20013256 (Registry Identifier: Regional Scientific Ethics Committee)
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 Diabetes; Hypoglycemia; Dasiglucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — dasiglucagon; Carbohydrates; Glucose

STUDY DESIGN:
Intervention Model Description: Single-blinded, randomized (using blocks of 3/6 and stratification by treatment modality), three-arm crossover study
Who Masked: Participant
Masking Description: Partially single-blinded (oral carbohydrate administration will not be blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 80 µg s.c. dasiglucagon (Experimental): 80 µg of dasiglucagon will be administered subcutaneously when plasma glucose levels reach 4.5 mmol/l
  Interventions: Drug: Dasiglucagon
- 120 µg s.c. dasiglucagon (Experimental): 120 µg of dasiglucagon will be administered subcutaneously when plasma glucose levels reach 4.5 mmol/l
  Interventions: Drug: Dasiglucagon
- 15 g oral carbohydrate (dextrose tablets) (Active Comparator): 15 g of oral carbohydrate (dextrose tablets) will be administered when plasma glucose levels reach 4.5 mmol/l
  Interventions: Other: Carbohydrate (dextrose tablets)

INTERVENTIONS:
Drug: Dasiglucagon — Abdominal s.c. administration
  Arms: 120 µg s.c. dasiglucagon; 80 µg s.c. dasiglucagon
Other: Carbohydrate (dextrose tablets) — Oral administration
  Arms: 15 g oral carbohydrate (dextrose tablets)

SUMMARY:
The aim of the study is to compare the efficacy of low-dose dasiglucagon (Zealand Pharma, Denmark) to oral carbohydrate consumption for prevention of s.c. insulin-induced hypoglycemia in CSII- and MDI-treated people with type 1 diabetes.

DETAILED DESCRIPTION:
Near-normalization of blood glucose levels through intensive insulin therapy has shown to reduce the risk of diabetes late complications, but the approach is associated with two major side effects: hypoglycemia and weight gain. Although management of hypoglycemia through oral carbohydrate consumption is generally effective, the approach can lead to excessive carbohydrate intake and cause rebound hyperglycemia. It has previously been demonstrated that subcutaneous (s.c.) low-dose glucagon can be utilized to effectively treat mild hypoglycemia in people with type 1 diabetes. However, the instability in aqueous solution of currently available glucagon and the need for reconstitution with sterile water immediately prior to administration has limited its clinical role outside emergency settings. Due to the stability and ready-to-use formulation, dasiglucagon does not hold the limitations known for the currently available glucagon preparations.

The aim of this randomized, partially single-blinded, three-arm cross-over study is to compare the efficacy of low-dose dasiglucagon (80 and 120 μg) to oral carbohydrate (15 g) consumption for prevention of s.c. insulin-induced hypoglycemia in CSII- and MDI-treated people with type 1 diabetes. On each study visit (separated by ≥ 3 days), an initial insulin bolus will be administered (at t = 0) aiming for a plasma glucose (PG) level of 3.0 mmol/l. When reaching 4.5 mmol/l, the intervention (s.c. dasiglucagon or oral carbohydrates) will be administered (t-intervention = 0), whereafter PG will me monitored for an additional 180 min.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* Duration of T1D ≥ 3 years
* Use of CSII or MDI therapy for ≥ 6 months
* Current use of Novorapid (change from another fast-acting insulin to Novorapid prior to study initiation is allowed)
* HbA1c ≤ 8.0%
* Regular use of carbohydrate counting in the judgement of the investigator

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* History of allergy or intolerance to glucagon or glucagon-like products
* Patients with pheochromocytoma
* Clinically significant ECG abnormalities
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (sterilization, intrauterine device, contraceptive pill, patch or injection)
* Inability to understand the individual information and to give informed consent
* Current participation in another clinical trial that, in the judgment of the principle investigator, will compromise the results of the study or the safety of the subject
* Other concomitant medical or psychological condition that, according to the investigator's assessment, makes the individual unsuitable for study participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Difference between study visits in time (min) in hypoglycemia (plasma glucose < 3.9 mmol/l) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)

SECONDARY OUTCOMES:
Difference between study visits in incidence rate of hypoglycemia (plasma glucose < 3.9 mmol/l) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in incidence rate of level 2 hypoglycemia (plasma glucose < 3.0 mmol/l) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in incidence rate of rebound hyperglycemia (plasma glucose > 10 mmol/l) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in nadir plasma glucose concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in peak plasma glucose concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in incremental peak in plasma glucose concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in mean plasma glucose concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time (min) from intervention to first increase in plasma glucose concentration of 1.1 mmol/l | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in plasma glucose Area Under the Curve (AUC) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time (min) to peak plasma glucose concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time (min) in range (plasma glucose ≥ 3.9 mmol/l and 10.0 mmol/l) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time (min) in hyperglycemia (plasma glucose > 10 mmol/l) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time (%) in hypoglycemia (plasma glucose < 3.9 mmol/l) (per protocol) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in incidence rate of rescue carbohydrate administration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time (min) to rescue carbohydrate administration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in plasma dasiglucagon Area Under the Curve (AUC) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in peak plasma dasiglucagon concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in time to peak plasma dasiglucagon concentration from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in serum insulin concentration at visit start (t = 0) and immediately before administration of the intervention (t-intervention = 0) | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in serum insulin AUC from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in dose (units) of insulin bolus at study start (t = 0) | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in change in Edinburgh Hypoglycemia Symptoms Scale (EHSS) from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in change in visual analogue scale (VAS) for nausea, headache, stomach ache, injection site pain, palpitations and hunger from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)
Difference between study visits in incidence rate of vomiting from 0-180 minutes post-intervention | Study visit 1 (day 1), study visit 2 (estimated day 4) and study visit 3 (estimated day 7)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Laugesen, MD, Principal Investigator — MD, PhD Candidate
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laugesen C, Ranjan AG, Schmidt S, Norgaard K. Low-Dose Dasiglucagon Versus Oral Glucose for Prevention of Insulin-Induced Hypoglycemia in People With Type 1 Diabetes: A Phase 2, Randomized, Three-Arm Crossover Study. Diabetes Care. 2022 Jun 2;45(6):1391-1399. doi: 10.2337/dc21-2304. PMID 35475907